CLINICAL TRIAL: NCT04246853
Title: Effects of Non Invasive Brain Stimulation on Experimental Pain
Brief Title: Effects of Non Invasive Brain Stimulation During Prolonged Experimental Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Luisina Gregoret, Biomedical engineer, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: N-20180092
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Pain; Prolonged Experimental Pain
MeSH Terms: conditions — Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The current studies have a randomized, parallel, sham-controlled and double-blinded design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinding is performed by a third-party which is not part of the research group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS of the resting state motor network (Active Comparator): The active comparator is the Active tDCS group. The active tDCS will target the resting-state motor network and will apply a distributed direct current during the whole session. (The TIME during the direct current is applied is the only difference with Sham tDCS) Each tDCS session lasts 20 minutes and applies a total current of 4mA.
  Interventions: Device: Transcranial direct current stimulation (tDCS) of the resting state motor network
- Sham tDCS of the resting state motor network (Sham Comparator): This study has a parallel design and 2 groups: Active tDCS and Sham tDCS. Sham tDCS applies a standard sham protocol consisting of ramping up and down during 30 seconds at the beginning and at the end of each tDCS session. Each tDCS session lasts 20 minutes and applies a total current of 4mA.
  Interventions: Device: Transcranial direct current stimulation (tDCS) of the resting state motor network

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) of the resting state motor network — Transcranial direct current stimulation (tDCS) delivers a low intensity current of up to 4 mA per session through small and circular shaped electrodes applied over the scalp. This induces a weak but focal electrical field that may modify the excitability of the underlying cortical target in a polarity and activity dependent fashion.

SUMMARY:
Non invasive brain stimulation (NIBS) of the primary motor cortex (M1) through transcranial direct current stimulation (tDCS) has been widely investigated in research and clinical settings in order to modulate brain plasticity and improve clinical pain. Interestingly, newly developed paradigms i.e. tDCS of the resting state motor network have proved higher modulatory effects in terms of corticospinal excitability when compared to traditional M1 tDCS.

However, little is known about the effects of tDCS on the frequency changes of alpha oscillations (alpha peaks).

Interestingly, previous studies show a correlation between reduced frequencies of alpha peaks during 1-hour experimental pain in comparison to baseline.

The present study aims to investigate the effects of tDCS of the resting state motor network on the frequency and power of alpha peaks during prolonged experimental pain during 24 hours.

DETAILED DESCRIPTION:
There is evidence that chronic pain alters the frequency of alpha peaks. Specifically, recent studies showed a correlation between decreased frequency of alpha peaks and perceived pain. Furthermore, a correlation was found between high pain sensitivity and slower alpha oscillations during prolonged pain during 1 hour.

To date, the effects of prolonged experimental pain during 24 hours on brain oscillations has not been explored. Moreover, it is unknown whether non invasive brain stimulation (NIBS) through transcranial direct current stimulation (tDCS) can revert these pain-related feature.

It is hypothesized that prolonged pain during 24 hours will reduce the frequency of alpha peaks and tDCS of the resting state motor network will revert it to baseline values.

Furthermore, it is thought that decreased frequency of alpha peaks will be correlated with perceived pain intensity on Day 1 (before receiving the first tDCS session).

ELIGIBILITY:
Inclusion Criteria:

* Right-handed healthy men and women in the age 21-50 years who speak and understand English

Exclusion Criteria:

* Lack of ability to cooperate
* History of chronic pain or current acute pain
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Present and previous neurologic, musculoskeletal or mental illnesses
* Chili allergies
* Current use of medications that may affect the trial
* Contraindications to rTMS application (history of epilepsy, metal implants in head or jaw, etc.)
* Failure to pass the questionnaire for tDCS

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Frequency of alpha peaks | 24 hours
  The frequency of alpha peaks will be extracted through electroencephalography (EEG) in the sensorimotor areas (Central-Parietal) of the brain. It is hypothesized that the frequency of alpha peaks will be reduced due to prolonged pain. It is expected that tDCS of the resting state motor network will revert the frequency to baseline values or even higher.
Perceived pain intensity | 24 hours
  Perceived pain intensity will be rated in a 0-10 Numerical rating scale (NRS): 0 no pain and 10 worst pain imaginable. Prolonged pain will increase perceived pain intensity. It is expected that active tDCS will not be able to reduce perceived pain intensity in comparison to sham tDCS.

SECONDARY OUTCOMES:
Amplitude of alpha peak | 24 hours
  Similar to the primary outcome, the amplitude of the alpha peak will be extracted through EEG in the sensorimotor area. It is expected that prolonged pain will be able to reduce the amplitude of alpha peaks and tDCS will increase it back to baseline values or even higher.
Power of alpha oscillations | 24 hours
  Spectral analysis will be performed on alpha activity and it is expected that this outcome will be reduced by prolonged pain and tDCS of the resting state motor network will be able to normalize it.

OTHER OUTCOMES:
Amplitude of Mu-oscillations during motor imagery | 24 hours
  Amplitude of Mu-oscillations will be extracted from EEG during motor imagery tasks (abduction-adduction of index finger). It is expected that prolonged pain and motor imagery will produce a desynchronization of Mu-oscillations and on the contrary active tDCS will be able to synchronize it back similar to pain-free state.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Nordylland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided